CLINICAL TRIAL: NCT04623099
Title: Pharmacogenetically-guided Escitalopram Treatment for Pediatric Anxiety: Aiming to Improve Safety and Efficacy (PrEcISE)
Acronym: PrEcISE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jeffrey Strawn, MD, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Strawn PrEcISE; R01HD099775 (NIH)
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Anxiety
Keywords: Kids; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: This randomized, controlled trial compares pharmacogenetically-guided and standard dosing of escitalopram in adolescents (12-17 years of age) with anxiety disorders. In this study, investigators will examine these two dosing strategies in terms of efficacy (Aim 1) and tolerability (Aim 2). Investigators will also evaluate the relationship between pharmacodynamic variables and treatment response.
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard dosing (Other): Patients randomized to standard dosing (std) will initiate escitalopram at 5 mg daily and will then increase to 20 mg/day at week 4.
  Interventions: Drug: Escitalopram
- Pharmacogenetically-guided escitalopram dosing (Experimental): Patients randomized to PGx-guided treatment, escitalopram titration will be based on CYP2C19 phenotype and predicted escitalopram exposure. In poor metabolizers (PM), escitalopram will be initiated at 5 mg daily and increased to 10 mg daily at week 4.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram is FDA-approved for the treatment of major depressive disorder (MDD) in adolescents (12-17 years of age) and is commonly prescribed for adolescents with anxiety disorders.
  Other Names: Lexapro

SUMMARY:
This double-blind, 12-week study will consist include132 anxious youth who are randomized (1:1) to standard or pharmacogenetically-guided escitalopram dosing. Block randomization (1:1) will be stratified by sex and metabolizer status.

DETAILED DESCRIPTION:
This randomized, controlled trial compares pharmacogenetically-guided and standard dosing of escitalopram in adolescents (12-17 years of age) with anxiety disorders. In this study, the investigators will examine these two dosing strategies in terms of efficacy (Aim 1) and tolerability (Aim 2).

The investigators propose to recruit 132 adolescents (age 12-17 years, inclusive) with generalized, separation and/or social anxiety disorder (pediatric anxiety trial).1 This will allow investigators to evaluate whether pharmacogenetically-guided escitalopram dosing improves efficacy and tolerability in outpatient adolescents aged 12-17 years with anxiety disorders. Eligible patients will be randomized to: (1) standard escitalopram dosing or (2) pharmacogenetically-guided dosing for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed assent and consent.
2. Patients, parent/guardian must be fluent in the English.
3. 12 to 17 years of age, inclusive, at Visit 1.
4. Patients must meet DSM-512 criteria for generalized, social and/or separation anxiety disorder, confirmed by the MINI-KID.
5. PARS score ≥15 at Visit 1 and Visit 2.
6. No initiation of psychotherapy within 8 weeks of screening (Visit 1). Current therapy much be stable for ≥2 months prior to baseline (Visit 2).
7. Clinical Global Impressions-Severity (CGI-S) score ≥4 at Visits 1 & 2.
8. Caregiver who is willing to consent to be responsible for safety monitoring of the patient, provide information about the patient's condition, oversee the administration of the investigational product.
9. No clinically significant abnormalities on physical examination and EKG.
10. Negative pregnancy test at Visit 1 in females.
11. Negative urine drug screen at Visit 1.
12. Sexually active patients must practice a reliable method of contraception that will continue for the duration of the study and for a minimum of 30 days following the end of study participation. Reliable methods of contraception are defined below; other forms of contraceptives (pharmacological and/or non-pharmacological) are not accepted:

    1. Surgical sterilization
    2. Oral contraceptives (e.g. estrogen-progestin combination or progestin)
    3. Transdermally-delivered contraceptives (e.g., Ortho-Evra), depot injections (e.g., Depo-Provera)
    4. Vaginal contraceptive ring (e.g., NuvaRing), contraceptive implants (e.g., Implanon, Norplant II/Jadelle)
    5. An intrauterine device
    6. Diaphragm plus condom. -

Exclusion Criteria:

1. Co-occurring DSM-5 mood disorder (except persistent depressive disorder, unspecified depressive disorder, provided that the primary diagnosis is an anxiety disorder), eating, bipolar or psychotic disorders.
2. A lifetime diagnosis of an intellectual disability.
3. A significant history of trauma exposure.
4. A history of SSRI treatment within 12 weeks of baseline or current treatment with a medication with psychiatric effects that requires >5 half-lives for washout History of non-response to >2 SSRIs.
5. Allergy, intolerance, non-response or hypersensitivity to escitalopram. Major neurological or medical illness or head trauma with ≥5 minutes loss of consciousness.
6. Alcohol or substance use disorder within the past 6 months (nicotine use is permitted).
7. Psychotherapy initiated within 8 weeks of screening (Visit 1), or plans to initiate/change therapy during the study.
8. Pregnant, breastfeeding, lactating, and/or planning to become pregnant during the study or within 30 days following the end of study participation.
9. Positive urine pregnancy test.
10. A positive urine drug screen.
11. Patient lives >90 minutes from UC or unable to attend follow-up visits. Suicide risk as determined by either: (1) any suicide attempt within the past 6 months and/or (2) significant risk at Visit 1 (Screening) or Visit 2 (Baseline), as judged by the Investigator.
12. QTc >450 in males or >460 in females (prolonged QTc based on American Heart Association recommendations for Standardization and Interpretation of the EKG
13. Patients who are unable to swallow capsules.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale severity score | Baseline to Week 12/Early Termination
  Change from Baseline in Pediatric Anxiety Rating Scale (PARS) severity score. The PARS is a clinician-rated instrument for assessing the severity of anxiety symptoms associated with common anxiety disorders in children and adolescents. The PARS score is derived by summing 5 of the 7 severity/impairment/interference items (2, 3, 5, 6, and 7)

SECONDARY OUTCOMES:
Tolerability-Activation | Baseline to Week 12/Early Termination
  Emergence of activation based on the Treatment-Emergent Activation and Suicidality Assessment Profile

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Strawn, MD, Principal Investigator — University of Cincinnati; Laura B Ramsey, PhD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- University of Cincinnati, Department of Psychiatry & Behavioral Neuroscience, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strawn JR, Poweleit EA, Mills JA, Schroeder HK, Neptune ZA, Specht AM, Farrow JE, Zhang X, Martin LJ, Ramsey LB. Pharmacogenetically Guided Escitalopram Treatment for Pediatric Anxiety Disorders: Protocol for a Double-Blind Randomized Trial. J Pers Med. 2021 Nov 12;11(11):1188. doi: 10.3390/jpm11111188. PMID 34834540